CLINICAL TRIAL: NCT01045837
Title: Effect of Addition of Short Course of Prednisolone to Gluten Free Diet and Gluten Free Diet Alone in the Recovery of Clinical, Histological and Immunological Features in Naive Adult Patients With Celiac Disease
Brief Title: Effect of Addition of Short Course of Prednisolone to Gluten Free Diet in Naive Celiac Disease Patients
Acronym: CD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Govind K Makharia, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Celiac-Prednisolone
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Celiac Disease
Keywords: Celiac disease, steroids, immunohistochemistry
MeSH Terms: conditions — Celiac Disease | interventions — Prednisolone; Diet, Gluten-Free; Steroids; Glutens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolone and Gluten free diet (Active Comparator): Gluten free diet and prednisolone in the dose of 1 mg/kg/d over a period of 4 weeks.
  Interventions: Drug: Prednisolone and Gluten free diet
- Gluten free diet (Placebo Comparator): Gluten free alone will be given in this group
  Interventions: Behavioral: Gluten free diet

INTERVENTIONS:
Drug: Prednisolone and Gluten free diet — Gluten free diet and Oral Prednisolone in a dose of 1 mg/ kg will be given for a period of 4 weeks, thereafter Gluten free diet alone will be continued
  Other Names: Steroids; Wysolone
  Arms: Prednisolone and Gluten free diet
Behavioral: Gluten free diet — Only gluten free diet will be given in this group
  Other Names: Gluten
  Arms: Gluten free diet

SUMMARY:
Withdrawal of gluten, the culprit antigen, is the definite treatment for celiac disease. Weeks to months after gluten withdrawal from the diet before the clinical manifestations, histological features start improving. Many of the adult patients are in the critical phase where even weeks may matter especially those in their adolescence where height growth has limited potential.

Suppression of immune system using a short course of steroid might retard the immune mediated destruction of the villi while the effect of gluten withdrawal sets in. Steroids are known to be effective in the management of refractory celiac disease. Therefore, the investigators hypothesized that addition of a short course of steroid to gluten free diet may enhance intestinal mucosal recovery and thus clinical manifestations

DETAILED DESCRIPTION:
Celiac disease is a chronic systemic autoimmune disorder induced by gluten proteins present in wheat, barley, and rye. Steroids affect proliferative responses of both B and T cells in vitro, and the production of lymphokines (migratory inhibitory factor) by cultured cells. Steroids inhibit the effect of gluten proteins through their action on elements of the immune system. Glucocorticoids are reserved for severely ill patients, who present with celiac crisis, gliadin shock, and refractory sprue. We hypothesized that addition of a short course of steroid to gluten free diet may enhance intestinal mucosal recovery and thus clinical manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Naïve patients with celiac disease (CD will be diagnosed as per revised European Society of Pediatric Gastroenterology and Nutrition criteria
* Both sexes
* Age>12 years

Exclusion Criteria:

* Partially treated celiac disease
* Co-existent systemic diseases
* HIV seropositive
* Seropositive with HBsAg , Anti HCV Ab
* Past H/O tuberculosis
* Evidence of active tuberculosis
* Unwilling patient

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having improvement in symptoms at 4 weeks | 4 weeks
Proportion of patients having improvement in histological improvement by at least one grade at 4 weeks | 4 weeks

SECONDARY OUTCOMES:
Proportion of patients showing normalization of histological abnormalities at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Govind Makharia, MD, DM, Principal Investigator — All India Institue of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Revised criteria for diagnosis of coeliac disease. Report of Working Group of European Society of Paediatric Gastroenterology and Nutrition. Arch Dis Child. 1990 Aug;65(8):909-11. doi: 10.1136/adc.65.8.909. No abstract available. PMID 2205160
- [Background] Katz AJ, Falchuk ZM, Strober W, Shwachman H. Gluten-sensitive enteropathy. Inhibition by cortisol of the effect of gluten protein in vitro. N Engl J Med. 1976 Jul 15;295(3):131-5. doi: 10.1056/NEJM197607152950303. PMID 1272329
- [Background] Mitchison HC, al Mardini H, Gillespie S, Laker M, Zaitoun A, Record CO. A pilot study of fluticasone propionate in untreated coeliac disease. Gut. 1991 Mar;32(3):260-5. doi: 10.1136/gut.32.3.260. PMID 1901562
- [Background] Balow JE, Rosenthal AS. Glucocorticoid suppression of macrophage migration inhibitory factor. J Exp Med. 1973 Apr 1;137(4):1031-41. doi: 10.1084/jem.137.4.1031. PMID 4693151
- [Background] Cellier C, Delabesse E, Helmer C, Patey N, Matuchansky C, Jabri B, Macintyre E, Cerf-Bensussan N, Brousse N. Refractory sprue, coeliac disease, and enteropathy-associated T-cell lymphoma. French Coeliac Disease Study Group. Lancet. 2000 Jul 15;356(9225):203-8. doi: 10.1016/s0140-6736(00)02481-8. PMID 10963198
- [Background] Marsh MN. Gluten, major histocompatibility complex, and the small intestine. A molecular and immunobiologic approach to the spectrum of gluten sensitivity ('celiac sprue'). Gastroenterology. 1992 Jan;102(1):330-54. PMID 1727768
- [Derived] Shalimar, Das P, Sreenivas V, Datta Gupta S, Panda SK, Makharia GK. Effect of addition of short course of prednisolone to gluten-free diet on mucosal epithelial cell regeneration and apoptosis in celiac disease: a pilot randomized controlled trial. Dig Dis Sci. 2012 Dec;57(12):3116-25. doi: 10.1007/s10620-012-2294-1. Epub 2012 Jun 30. PMID 22752636